CLINICAL TRIAL: NCT00377091
Title: Pilot Pharmacoeconomic Evaluation of Fondaparinux Treatment of Pulmonary Embolism (PE) Compared to Treatment With Unfractionated Heparin
Brief Title: Is Using Fondaparinux (Blood Thinner) to Treat Lung Clot Cheaper Than Traditional Therapy
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: Study pulled due to a grant disagreement between the U of M and SMDC
Sponsor: University of Minnesota (Other)
Collaborators: GlaxoSmithKline (Industry)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0510M76771
Record Dates: First submitted 2006-09-13; First posted 2006-09-15 (Estimated); Last update posted 2013-05-30 (Estimated); Status verified 2013-05

CONDITIONS: Pulmonary Embolism
Keywords: pulmonary embolism; venous thromboembolism; pharmacoeconomic; heparin; unfractionated heparin; fondaparinux; length of stay; costs; bleeding; thrombosis
MeSH Terms: conditions — Pulmonary Embolism; Venous Thromboembolism; Hemorrhage; Thrombosis | interventions — Fondaparinux

INTERVENTIONS:
Drug: Fondaparinux

SUMMARY:
This study compares two blood thinners which are both accepted standard cares, fondaparinux and unfractionated heparin (UFH). These drugs are used to prevent the growth of existing blood clots and formation of additional blood clots in patients with pulmonary embolism (a blood clot in the lung) as they are beginning to take warfarin (another standard care blood thinner). Patients will be invited to participate because they have been diagnosed with a pulmonary embolism, require anticoagulation therapy (treatment with a blood thinner), and are currently hospitalized.

The purpose of this study is to determine if patients treated with fondaparinux will have shorter hospital stays and lower costs of treatment while in the hospital than similar patients receiving a different standard care with UFH. Fondaparinux is already approved by the FDA for use in patients with pulmonary embolism, for both inpatient and outpatient care, as long as treatment is begun with warfarin while they are hospitalized. It is therefore not an experimental treatment. The study is being conducted to determine which FDA approved treatment is the best practice for hospital treatment of pulmonary embolism. The study will also examine the safety and effectiveness of fondaparinux in local use.

DETAILED DESCRIPTION:
Research Question

This study is being conducted to determine if treatment of pulmonary embolism (PE) with fondaparinux will decrease the length of stay and hospital costs of therapy while maintaining safety and efficacy, when compared to unfractionated heparin (UFH). Primary research questions: Determine if PE treatment utilizing fondaparinux will reduce the inpatient length of stay (LOS) and costs of hospital care to St. Mary's Duluth Clinic Health System (SMDC), when compared to a matched group of patients treated with UFH as standard care, during the same time period. Secondary research questions: Determine if bleeding and recurrent thrombosis rates are similar between the fondaparinux cohort and the UFH matched control group.

Specific Aims

1. Enroll 30 St. Mary's Medical Center (SMMC, an affiliate of SMDC) patients into the treatment cohort, utilizing fondaparinux as their primary immediate antithrombin therapy, while warfarin is being titrated to therapeutic effect.
2. Retrospectively identify a matched control group of 30 PE patients, treated with UFH as standard care, during the same period of time.
3. Determine the LOS and costs of inpatient care on a standardized scale for both the treatment cohort and the control group.
4. Perform a retrospective review of patients' medical records for the 3 months after the initial pulmonary embolism, to determine the rates of:

4a. repeat venous thromboembolism events (VTE) 4b. bleeding events

ELIGIBILITY:
Inclusion Criteria:

1. Patients 18 years of age or older who present with acute symptomatic pulmonary embolism and who require antithrombotic therapy
2. Diagnostic confirmation based on the following criteria

   1. intraluminal filling defect on spiral computed tomography (CT) or pulmonary angiography
   2. a high-probability ventilation-perfusion lung scan, or a nondiagnostic lung scan with documentation of deep-vein thrombosis, either by compression ultrasonography or by venography.
3. Primary outpatient MD of record is an SMDC MD or patient did not have an outpatient MD when this event occurred.
4. For the matched control (UFH) cohort only: unfractionated heparin utilized for initial antithrombotic therapy. (LMWH use is allowed initially in the fondaparinux arm.) Patient willingness to have fondaparinux injections administered as an outpatient by themselves, family members, or other caregivers.

Exclusion Criteria:

1. Patients will be ineligible for the study if they had received therapeutic doses of UFH or LMWH or oral anticoagulants for more than 24 hours;
2. Patient required thrombolysis, embolectomy, or a vena cava filter;
3. Anticoagulant therapy was contraindicated - for example, because of active bleeding or thrombocytopenia (a platelet count below 100,000 per cubic millimeter).
4. Patients are ineligible if they had an estimated creatinine clearance < 30 mL/min.
5. Uncontrolled hypertension (systolic blood pressure greater than 180 mm Hg or diastolic blood pressure greater than 110 mm Hg);
6. Pregnancy
7. Physician has estimated the life expectancy to be less than three months.
8. Patients weighing > 150 kg
9. Indwelling epidural catheter
10. Inability to give informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2007-06; Primary Completion 2007-11 (Actual); Study Completion 2007-11 (Actual)

PRIMARY OUTCOMES:
Primary endpoints: The primary end-points will be determining if the utilization of fondaparinux to treat PE in the inpatient setting will reduce length of stay and hospital treatment costs, when compared to a UFH matched control group.

SECONDARY OUTCOMES:
Secondary endpoints: The secondary end-points will be to determine if bleeding and recurrent thrombosis rates are similar between the fondaparinux cohort and the UFH matched control group.

CONTACTS AND LOCATIONS:
Overall Officials: Michael P. Gulseth, Pharm. D., Principal Investigator — University of Minnesota
Locations (1):
- St. Mary's Medical Center, Duluth, Minnesota, United States